CLINICAL TRIAL: NCT06900673
Title: Reducing Disparities in Access to Evidence-Based Services for ADHD Through Technology
Brief Title: Reducing Disparities in Access to Evidence-Based Services for Attention Deficit Hyperactivity Disorder (ADHD) Through Technology
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Francisco (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2024-0193; U54MD012397 (NIH)
Record Dates: First submitted 2025-03-18; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Control Condition; Intervention Condition
Keywords: ADHD; digital health technology; school mental health; health equity; child mental health
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Business As Usual (No Intervention): Students in the control condition will receive the usual services their schools provide to students with or at risk for ADHD in grades 2-5.
- Collaborative Life Skills (Experimental): Student, parents, and teachers in the intervention condition will receive the digitally adapted Collaborative Life Skills program.
  Interventions: Behavioral: Collaborative Life Skills

INTERVENTIONS:
Behavioral: Collaborative Life Skills — Student, parents, and teachers in the intervention condition will receive the digitally adapted Collaborative Life Skills program.
  Arms: Collaborative Life Skills

SUMMARY:
This project aims to develop an adaptation of the Collaborative Life Skills Program (CLS) that will be supported by mHealth technology. CLS is an evidence-based intervention for 2nd-5th grade children with ADHD that is delivered in schools through coordinated efforts among school mental health providers, teachers, and parents. School mental health providers are trained to coordinate evidence-based teacher- (i.e., Daily Behavioral Report Card) and parent-mediated (i.e., Behavioral Parent Training) behavioral interventions, and lead child social and organizational skills training groups. The adapted intervention, which integrates mHealth technology (CLS-M), will improve the usability, feasibility, and acceptability of CLS in schools with limited resources serving children from low-socioeconomic status (SES) and ethnic/racial minority (ERM) backgrounds, reducing disparities in access to evidence-based ADHD interventions in these populations. Barriers to service use in schools where low-SES and ERM families are most likely to receive services include logistical constraints (e.g., time, transportation, childcare, work schedules), perceptual barriers (e.g., cultural mistrust, stigma, perceived efficacy), and insufficient resources (e.g., staff, time, consultation support). Building on prior research, the investigators will develop and test a fully functional web-based mHealth application to support CLS-M that includes an integrated user portal for school mental health providers, teachers, and parents. The application will also include separate interfaces that support key features to facilitate each person's role in CLS implementation at school or at home, such as access to shared information about child assessments, goals, and automatically generated graphs of child Daily Behavioral Report Card performance. Messaging features will facilitate communication among school mental health providers, parents, and teachers, and calendar features that integrate with third- party calendar applications (e.g., Google Calendar) will facilitate scheduling, meeting tracking, and sharing links to third-party videoconferencing applications (e.g., Zoom). Based on stakeholder feedback from school administrators, school mental health providers, teachers, and parents, the investigators will work with mobile application developers to design a fully functional web-based mHealth application prototype to support the CLS-M protocol. the investigators will then test and refine the prototype through a series of individual usability tests and an open feasibility trial. the investigators will also collect formative data from stakeholders in rural schools in Imperial County to inform future research on adapting CLS-M for low-SES and ERM families served in this setting. Finally, the investigators will conduct a Hybrid Type I cluster randomized trial in 24 schools in a large urban school district, to evaluate whether CLS-M results in acceptable implementation outcomes and improved child outcomes in comparison to usual school services. The specific aims are to 1) Develop CLS-M and test its usability, feasibility, and acceptability among key stakeholders; 2) Collect formative data to inform future CLS-M adaptations for families living in rural settings; and 3) Evaluate CLS-M implementation and impact on child outcomes relative to typical school services.

DETAILED DESCRIPTION:
The proposed pilot project aims to extend the reach of evidence-based behavioral intervention services for children from low-SES and ERM families by developing the first school-based after-school intervention model for elementary school children with ADHD and enhancing it with mobile health (mHealth) technology. In partnership with an urban elementary school, the investigators will recruit panels of key opinion leaders representing five stakeholder groups, including teachers, school mental health professionals, after-school staff, parents, and children with ADHD to participate in a series of three focus groups that aim to:

Aim 1: Assess the existing resources, organizational capacity, and unmet needs of low-SES and ERM children with ADHD at the school. Focus groups will be conducted with each stakeholder panel to identify the service capacity and unmet needs of children with ADHD. A logic model of the problem will be developed to inform the identification of existing evidence-based interventions and mHealth solutions that could fit the context.

Aim 2: Adapt existing interventions and design mock mHealth application prototypes. Intervention models and mHealth solutions will be presented to stakeholder panels in a second set of focus groups to solicit feedback about the perceived need for adaptations to the interventions and fit of the mHealth solutions with the needs, environment, conditions, capacity, and culture of the target school/population. Adaptations will be made the to intervention and mock mHealth examples based on stakeholder feedback will produce an intervention model prototypes.

Aim 3: Evaluate the perceived usability, acceptability and feasibility of the intervention model and mock mHealth prototypes. A third set of focus groups with stakeholder panels will assess their perceptions of the intervention model and mock mHealth prototypes. Usability testing of the mHealth prototypes will be conducted with three members of each panel to identify design issues, assess task completion, and solicit user feedback.

Impact: The findings of the present project will lay the foundation for a subsequent proposal for funding (e.g., R21, R34) to further develop the intervention materials and mHealth applications and evaluate their feasibility and initial impact in a pilot implementation trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants in study must be be teachers, parents of children with ADHD, and school mental health providers.
* Students will be identified by school staff and administrators, with whom the investigators have existing relationships.
* Caregivers/parents will be included if their students are:

  * Enrolled full-time in a participating elementary schools.
  * In a mainstream classroom for the majority of the school day
  * In 2nd- 5th grade
  * Are eligible for free or reduced lunch
* Parents must also live with the identified child.

Exclusion Criteria:

• Parents are excluded from the study if their children have:

* Significant visual impairment
* Significant hearing impairment
* Severe language delay
* Psychosis
* Pervasive developmental disorder
* Global intellectual impairment.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Symptom Inventory-5 | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Parents and teachers will complete the Child and Adolescent Symptom Inventory-5 , which includes 78 items assessing DSM-5 symptoms of ADHD, ODD, CD, Mood, and Anxiety. It has demonstrated adequate reliability (rs = .66-.78) and internal consistency (αs = .90-.94).
Children's Organizational Skills Scales | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Parents and teachers will complete the Children's Organizational Skills Scales (COSS), which includes subscales assessing organizational skills, management of materials/supplies, and task planning skills (parent = 58 items, teacher = 35 items), with items rated on a 4-point scale. The parent and teacher versions both have excellent internal consistency (αs = .98 and .97, respectively), test-retest reliability (rs = .99 and .94, respectively), and evidence of structural, convergent, and discriminant validity.
Impairment Rating Scale | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Parents and teachers will report about students' functioning (e.g., academic, behavioral, peer, etc.) on the Impairment Rating Scale using a 6-point scale (0 = "needs no treatment" to 6 = "definitely requires treatment") with a rating greater than 2 suggests significant impairment requiring intervention.
Homework Problems Checklist | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Parents will complete the Homework Problems Checklist which consists of 20 items rated on a 4-point scale and has evidence of excellent internal consistency (α = .90-.92) to assess child problems related to homework.
Academic Competency Evaluation Scale | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Teachers will complete the Academic Enablers scale of the Academic Competency Evaluation Scale, which measures behaviors that support adaptive learning in the classroom. This subscale demonstrates excellent psychometric properties, including high test-retest reliability (r = .96) and internal consistency (α = .98) for children in grades 3-5.

SECONDARY OUTCOMES:
Alabama Parenting Questionnaire | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Parents will complete the Alabama Parenting Questionnaire (APQ), which consists of 42 parent-reported items and five subscales: involvement, positive parenting, monitoring, inconsistent discipline, and corporal punishment. The subscales have been validated using confirmatory factor analysis and have demonstrated evidence of reliability and validity.
Parent-Teacher Involvement Questionnaire | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  Parents and teachers will complete the Parent-Teacher Involvement Questionnaire (PTIQ) which consists of 47 items and six subscales: parent-teacher contact, parent involvement at school, quality of parent-teacher relationship, teacher's perception of the parent, parent involvement at home, and parent endorsement of school. The subscales have been validated using confirmatory factor analysis and have demonstrated evidence of reliability and validity.

OTHER OUTCOMES:
Intervention Fidelity | Completed in-vivo during during weekly parent and student group during the 8-week intervention
  Fidelity monitoring observation checklists will be adapted in Year 1 from those previously developed for CLS to measure fidelity of SMHP training in CLS-M, as well as SMHP implementation of each component of the CLS-M. A separate measure of SMHP competence in executing the treatment will be adapted from the CLS Implementation Quality Form used in previous trials, which will be completed by the trainer after each "live" observation. Items assess clarity of skill presentation, thoroughness of homework review, use of practical examples, and effectiveness of handout review rated by the trainer on a 1- 5 scale (from 1 = not at all to 5 = most). The child-group version includes items such as use of effective commands, prompts and praise, and clarity of skill presentation rated by the trainer on a 1-5 scale (from 1 = not at all to 5 = most). An independent research team member (blinded to group assignment) will rate 15% of sessions to estimate inter-rater reliability
Parent Strategy Use Questionnaire | Completed each week during the 8-week intervention directly following the parent group intervention
  Each week, parents will complete the 5-item Parent Strategy Use Questionnaire, a scale used in previous CLS trials to assess the frequency (rated on a 5-point scale) of parent's self-rated use of specific strategies taught during the previous Behavioral Parent Training sessions over the past week.
Daily Behavioral Report Card Completion | Completed throughout each day during the 8-week intervention period
  The proportion of school days the school and home Daily Behavioral Report Cards (DBRCs) were implemented each week will be calculated based on the number of completed DBRCs, divided by the overall count of possible days during the week, as the investigators have done in previous trials.
  School holidays (coded from the online student calendar for each school), child absence, special school events/field trips and substitute teacher days (when noted on the DBRC) will not be included in the overall count of possible school days during the week.
Feasibility Rating Scale | Completed each week during the 8-week intervention directly following weekly intervention groups
  SMHPs, teachers, and parents will complete the Feasibility Rating Scale, which consists of items regarding the amount of time required to participate in the intervention, the level of effort needed to identify and enroll children in the program, the availability of physical space needed to run in-person groups, etc. The investigators will query SMHPs weekly about CLS-M demands on their time, with specific questions regarding their use of the mHealth tool. At post-intervention, SMHPs, teachers, and parents will be queried about factors that might affect CLS-M implementation, including school resources needed for CLS-M (e.g., staff, space, materials, technology), teacher and parent involvement, logistical barriers (e.g., parent work schedules, childcare), and competing responsibilities and school needs.
Intervention Satisfaction | Completed each week during the 8-week intervention directly following weekly intervention groups
  SMHPs, parents, teachers, and children will complete satisfaction measures adapted from those used in previous CLS trials. Parents, teachers, and children in the CLS-M group will complete satisfaction questionnaires after each session pertaining to the content (e.g., usefulness, clarity, engagement, and applicability of topics/activities) and format (e.g., videoconferencing features) of that session, as well as their perceptions of specific features and components of the tool (e.g., data visualization formats, skills content, behavior/reinforcement tracking). The participants will also complete questionnaires at post-treatment and follow-up about their overall satisfaction with CLS-M, the mHealth tool, and their perceived level of child improvement. All items will be rated on a 5-point scale (1 = not at all, 5 = great deal). SMHPs will also complete satisfaction measures weekly and at post-treatment and follow-up regarding their perceptions of CLS-M features.
System Usability Scale | Following usability testing; the week after the end of the 8-week intervention
  Parents, teachers, and SMHPs will complete the System Usability Scale (SUS; Lewis & Sauro, 2009), a 10-item technology-agnostic scale assessing technology product usability. SUS scores above 80 indicating good usability (Lewis & Sauro, 2018). The SUS has high internal consistency (α = .91) and high convergent validity with a separate rating of usability and user satisfaction (r = .8). The SUS will be completed by SMHPs, teachers, and parents following usability tests, halfway through and at the end of the open trial, and at the post-intervention assessment of the cluster randomized trial.
Services for Children and Adolescents Parent Interview | Screening, Baseline, the week after the end of the 8-week intervention, and follow-up approximately 2 months after the subsequent school year starts.
  The Services for Children and Adolescents Parent Interview assesses children's use of mental health services (including medication), primary care services, school-based interventions, and community services. In previous CLS trials, the investigators have included questions about specific CLS components (e.g., DBRC, child skills training, parenting groups).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villodas, PhD, Principal Investigator — Department of Psychology, College of Sciences, San Diego State University; Linda Pfiffner, PhD, Principal Investigator — Department of Psychiatry, School of Medicine, University of California San Francisco
Locations (1):
- San Diego State University HealthLINK Center for Transdisciplinary Health Disparities Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No